CLINICAL TRIAL: NCT02470130
Title: Effect of a Debriefing Conversational Relaxation on Memorization of Critical Key Points in Resident High Fidelity Simulation Education Program
Brief Title: Relaxation Before Debriefing and Memorization in High Fidelity Simulation in Healthcare
Acronym: RELAXSIMHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, MD, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CLESS 2014
Record Dates: First submitted 2015-05-20; First posted 2015-06-12 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-07

CONDITIONS: Anxiety
Keywords: simulation; anxiety; debriefing; memorization
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- relax actor (Active Comparator): actor during simulation and relaxation before debriefing
  Interventions: Behavioral: relaxation
- no relax actor (No Intervention): actor during simulation and no relaxation before debriefing
- relax observer (Active Comparator): observer during simulation and relaxation before debriefing
  Interventions: Behavioral: relaxation
- no relax observer (No Intervention): observer during simulation and no relaxation before debriefing

INTERVENTIONS:
Behavioral: relaxation — 5 min of conversational relaxation red by one of the instructor between simulation and debriefing
  Arms: relax actor; relax observer

SUMMARY:
Resident in advanced medical training participated to high fidelity simulation education program in Lyon. Alternatively 1 or 2 resident act during a scenario while the others observe in a teletransmission closeby room. Debriefing follows the critical scenario in witch resident are involved. The investigators are testing the effects of five minute of conversational relaxation before the debriefing on the anxiety level and memorization of key points each scénario on participant and observer.

DETAILED DESCRIPTION:
Resident in advanced medical training participated to high fidelity simulation education program in Lyon. This is part of a curriculum and each year they go throw a specific simulation session in groups of 3 to 8 residents with same specific thematic education goals. 3 to 4 differents scénario are run every simulation session during 4 to 5 hours, every day 2 similar session are run with 2 different groups of same level residents. Alternatively 1 or 2 resident act during a scenario while the others observe in a teletransmission room. Debriefing follows the critical scenario in witch resident are involved. The investigators are testing the effects of five minute of conversational relaxation before the debriefing on the anxiety level and memorization of key points each scénario on participant and observer. Relaxation is done reading a text outloud by an instructor before the debriefing. Each scenario is run in the morning and the afternoon and alternatively have relaxation or not. evaluation is done on participant of the scenario and resident observer of the situation. The Investigators ask participant for demographic data, anxiety scale test, multiple anxiety visual analogic scale. At the end of every scenario 5 clinical key point of teh scenario are exposed. At 3 month the investigators call back every participant to ask them to remember these 5 points for the scenario they were involved in and one of the other they observed.

ELIGIBILITY:
Inclusion Criteria:

* every resident going to a scheduled simulation session part of the normal education program of the residency.

Exclusion Criteria:

* no consent, or consent deleted

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
memorization of the active scenario | 3 month
  5 key points for the resolution of the scenario, 1 point per key points recalled by the participant, metrics from 0 to 5.

SECONDARY OUTCOMES:
anxiety | min 1
  visual analog scale : metrics from 0 to 100 mm
debriefing | min 1
  score of quality of the debriefing questionnaire of 6 items quoted, total score from 25 to 175
observing | min 1
  visual analog scale : metrics from 0 to 100 mm
memorization of the passive scenario | 3 month
  5 key points for the resolution of the scenario, 1 point per key points recalled by the participant, metrics from 0 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: jean jacques Lehot, PHD, Study Chair — HCL
Locations (1):
- CLESS, Lyon, Auvergne-Rhône-Alpes, France